CLINICAL TRIAL: NCT02259816
Title: Pharmacokinetics of Repeated Oral Doses of 80 mg Telmisartan (Micardis®) at Steady State Alone and in Combination With Repeated Oral Doses of Amlodipine 10 mg (Norvasc®) at Steady State. A Two-way Crossover, Open, Randomised Design Study
Brief Title: Pharmacokinetics of Telmisartan Alone and in Combination With Amlodipine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1235.2
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Amlodipine

ARMS (2):
- Telmisartan (Active Comparator)
  Interventions: Drug: Telmisartan
- Telmisartan and amlodipine (Experimental)
  Interventions: Drug: Telmisartan; Drug: Amlodipine

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®
Drug: Amlodipine
  Other Names: Norvasc®
  Arms: Telmisartan and amlodipine

SUMMARY:
Study to investigate the steady state pharmacokinetics of 80 mg telmisartan alone and in combination with repeated doses of 10 mg amlodipine

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥18 and Age ≤50 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
10. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/corrected QT interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
11. Participation in another trial with an investigational drug within two months prior to administration or during the trial
12. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
13. Inability to refrain from smoking on trial days
14. Alcohol abuse (more than 60 g/day)
15. Drug abuse
16. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
17. Excessive physical activities (within one week prior to administration or during the trial)
18. Any laboratory value outside the reference range that is of clinical relevance
19. Inability to comply with dietary regimen of trial site
20. Any history of relevant low blood pressure
21. Supine blood pressure at screening of systolic <110 mm Hg and/or diastolic <60 mm Hg
22. History of urticaria

    For female subjects:
23. Pregnancy or planning to become pregnant within 2 months of study completion
24. Positive pregnancy test
25. No adequate contraception e.g. sterilisation, intrauterine device, have not been using a barrier method of contraception for at least 3 months prior to participation in the study
26. Are not willing or are unable to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and up to 2 months after completion/termination of the trial
27. Chronic use of oral contraception or hormone replacement containing ethinyl estradiol as the only method of contraception
28. Partner is unwilling to use condoms
29. Lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of telmisartan in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | up to 15 days after first administration of study drug
Maximum measured concentration of telmisartan in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | up to 15 days after first administration of study drug

SECONDARY OUTCOMES:
AUCτ,ss for amlodipine | up to 15 days after first administration of study drug
Cmax,ss for amlodipine | up to 15 days after first administration of study drug
Maximum measured concentration of the analyte in plasma (Cmax) | up to 12 hours after first administration of study drug
Time from dosing to maximum measured concentration on plasma (tmax) | up to 12 hours after first administration of study drug
Area under the plasma concentration-time curve over a uniform dosing interval τ after administration of the first dose; corresponds to AUC0-24h (AUCτ,1) | up to 12 hours after first administration of study drug
Pre-dose concentration of the analyte in plasma immediately before the administration of the next dose N (Cpre,N) | pre-dose on days 2-9
Time from last dosing to the maximum concentration of the analyte in plasma at steady state (tmax,ss) | up to 144 hours after last administration of study drug
Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | up to 144 hours after last administration of study drug
Terminal rate constant in plasma at steady state (λz,ss) | up to 144 hours after last administration of study drug
Terminal half-life of the analyte in plasma at steady state (t1/2, ss) | up to 144 hours after last administration of study drug
Mean residence time of the analyte in the body at steady state after oral administration (MRTpo,ss) | up to 144 hours after last administration of study drug
Apparent clearance of the analyte in plasma at steady state after extravascular multiple dose administration (CL/F,ss) | up to 144 hours after last administration of study drug
Apparent volume of distribution of the analyte in plasma at steady state after extravascular multiple dose administration (Vz/F,ss) | up to 144 hours after last administration of study drug
Accumulation ratio of the analyte in plasma based on AUC over a uniform dosing interval after the first and last doses (RA, AUC) | up to 15 days after first administration of study drug
Accumulation ratio of the analyte in plasma based on Cmax over a uniform dosing interval after the last and first doses (RA,Cmax) | up to 15 days after first administration of study drug
Number of subjects with adverse events | up to 80 days
Assessment of tolerability by investigator on a 4-point scale | within 14 days after last trial procedure